CLINICAL TRIAL: NCT06729684
Title: Development and Validation of Personalized Digital Healthcare Technology and Service Model for the Management and Recovery of Side Effects of Treatment in Breast Cancer Survivors
Brief Title: Development and Validation of a Personalized Digital Healthcare Model for Managing Side Effects in Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SMC 2023-10-048-010; HA23C0423 (Other: National Cancer Center (NCC))
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Survivorship; Breast Cancer; Digital Health
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Conventional Treatment) (No Intervention): * breast cancer surgery with CTx/RTx/HTx
  * brochure training
- intervention (digital health) (Experimental): * breast cancer surgery with CTx/RTx/HTx
  * brochure training
  * add digital health (application + smartwatch)
  Interventions: Device: digital health (application and smartwatch)

INTERVENTIONS:
Device: digital health (application and smartwatch) — The application allows users to conduct self-assessments for managing symptoms and side effects related to treatment. Based on the assessment results, it provides personalized self-management strategies. Additionally, users can access features for exercise, diet, and weight management.
  Arms: intervention (digital health)

SUMMARY:
The ultimate goal of this research and development is to develop personalized digital healthcare technologies and self-management strategies based on self-assessment results and evidence, for breast cancer survivors who require management and recovery from acute and chronic side effects related to various treatments (surgery, chemotherapy, radiation, hormone therapy, etc.). Additionally, the aim is to verify the clinical applicability and establish a service model to address the diverse unmet healthcare needs of breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have undergone surgery for Stage 1-2 breast cancer
* Individuals who have had a unilateral mastectomy
* Aged 18 years or older and under 65 years
* Possessing a smartphone with either an Android or iOS operating system
* Individuals who voluntarily decide to participate after receiving detailed information about the study and provide written consent

Exclusion Criteria:

* Individuals who have undergone mastectomy only and are not receiving chemotherapy, radiation, or hormone therapy
* Individuals with severe comorbidities (such as underlying diseases, neuromuscular disorders, cognitive or mental impairments, visual disabilities, etc.) that make it difficult to use the application or participate in the exercise intervention

Discontinuation Criteria

* Individuals who undergo delayed breast reconstruction surgery during the study period
* Individuals who develop severe complications or experience cancer metastasis or recurrence in other organs during the study period, leading to a change in treatment
* Occurrence of a major illness unrelated to study participation
* Failure to comply with the instructions of the study physician
* Situations where the participant voluntarily withdraws from the study or becomes unable to continue participating

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS29 | Baseline, Month 1, Month 3, Month 6
  Full Title: Patient-Reported Outcomes Measurement Information System Objective: health related quality of life Scoring System: Each item is rated on a scale of 1 to 5. Lower scores indicate better health for pain, depression, anxiety, and fatigue, while higher scores indicate better health for physical function, social roles, and activities, and sleep disorders.

SECONDARY OUTCOMES:
EQ-5D-5L | Baseline, Month 1, Month 3, Month 6
  Full Title: EuroQol 5-Dimension 5-level Objective: quality of life Scoring System: Each item is evaluated on a 5-point scale and weighted according to the country. EQ VAS evaluates data on a scale of 0-100, with a higher score indicating better health.
PRO-CTCAE | Month 1, Month 3, Month 6
  Full Title: Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events Objective: Clinical symptoms and adverse effects reported by patients Scoring System: Evaluate the frequency, severity, interference with daily activities, amount, and presence/absence of side effects over the past 7 days.
ICF (International Classification of Functioning, Disability, and Health) | Baseline, Month 1, Month 3, Month 6
  Full Title: International Classification of Functioning, Disability and Health Objective: function, activity and participant, environment
  Scoring System:
  A. Assess the 8 items of body functions, 8 items of activities and participation, and 8 items of environmental factors of the breast cancer ICF core set brief B. Body functions are assessed as 0 (no problems) - 4 (extreme problems), 9 (not applicable). Activities and participation are assessed as 0 (no difficulties) - 4 (extreme difficulties), 9 (not applicable). Environment is assessed as 0 (no barriers) - 4 (extreme barriers), +0 (no facilitating factors) - +4 (complete facilitating factors), 9 (not applicable).
Activity (step count) | Baseline, Month 1, Month 3, Month 6
  Objective: Number of steps taken in the past month Scoring System: Number of steps measured by mobile phone
TTM (Transtheoretical Model) | Baseline, Month 3, Month 6
  Full Title: The Transtheoretical Model staging Objective: behavior change stage
  Scoring System:
  A. Assess health behavior change on a 5-step scale B. (1) Before consideration: No intention to change problem behavior or adopt healthy behavior within the next 6 months, (2) Consideration: No specific plan but plan to take action within the next 6 months, (3) Preparation: Plan to take action within the next 30 days, (4) Action: In progress (less than 6 months), (5) Maintenance: In progress (more than 6 months) C. Check whether the change in the stage has occurred in a positive direction
OBQ-K | Baseline, Month 3, Month 6
  Full Title: Occupaitonal Balance Questionnaire Objective: occupational balance Scoring System: 13 items, 0-5 point scale. The score range is 0-65 points, and a higher score indicates greater work balance.
CBI-K | Baseline, Month 3, Month 6
  Full Title: Cancer Behavior Inventory version 3.0 - Korea Objective: Measuring self-efficacy for coping behaviors that can be taken during cancer treatment
  Scoring System:
  A. Consists of 7 subscales (27 items): Maintaining activity and independence (4 items), Seeking and understanding medical information (4 items), Managing stress and pain (4 items), Managing side effects (4 items), Accepting cancer/maintaining a positive attitude (4 items), Finding social support (3 items), Using spiritual coping methods (4 items) B. Rating on a 7-point scale. A higher score indicates a higher self-efficacy for overcoming cancer.
body composition (inbody) | Baseline, Month 1, Month 3, Month 6
  Weight: kg BMI(Body mass index): kg/m^2 SMI(Appendicular Skeletal Muscle Mass Index): kg/m^2

OTHER OUTCOMES:
SUS | Month 6
  Full Title: System Usability Scale Objective: System Usability
  Scoring System:
  A. 10 questions, 5-point scale B. Total = ((sum of odd questions - 5) + (25 - sum of even questions)) * 2.5 C. Score range is 0-100, and the benchmark is known to be 68 points.
satisfaction survey | Month 6
  Objective: Check app satisfaction and suggestions/issues
  Scoring system:
  A. Self-administered questionnaire b. Use a semi-structured survey to assess app satisfaction and gather suggestions/issues.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Republic of Korea, South Korea

IPD SHARING:
Plan to Share IPD: No